CLINICAL TRIAL: NCT05808608
Title: A Study of AK104 Plus Axitinib in Advanced/Metastatic Special Pathological Subtypes of Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hao Zeng (Other)
Responsible Party: Sponsor-Investigator, Hao Zeng, professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104AXI-ssRCC
Record Dates: First submitted 2023-03-23; First posted 2023-04-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Renal Cell Carcinoma; First-line Treatment; Non Clear Cell Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination treatment group (Experimental): Subjects in this group will receive AK104 (RP2D, administered intravenously) plus Axitinib 5 mg bid, administered orally.
  Interventions: Drug: AK104; Drug: Axitinib

INTERVENTIONS:
Drug: AK104 — Anti-PD-1/CTLA-4 bi-specific antibody drug; RP2D intravenously (IV)
Drug: Axitinib — An oral, small molecule, TKI selective for VEGFRs; 5mg bid orally

SUMMARY:
This is a Phase Ib/II, open-label, single arm trial to evaluate the efficacy and safety of AK104 in combination with axitinib as a first-line treatment for advanced/metastatic special pathological subtypes of renal cell carcinoma (ssRCC). Subjects will receive AK104 plus axitinib until disease progression, development of unacceptable toxic effects, death, a decision by the physician or patient to withdraw from the trial. The primary endpoint is ORR and PFS per RECIST v1.1 and imRECIST as assessed by investigators.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18, ≤75;
2. histology characteristics accord with special pathological subtypes of RCC: papillary renal cell carcinoma, chromophobic cell carcinoma, TFE3 rearrangement renal cell carcinoma, FH-deficient renal cell carcinoma, collecting duct carcinoma, medullary carcinoma, sarcomatoid carcinoma (>10%), unclassified renal cell carcinoma ;
3. metastatic renal cell carcinoma (TNM IV stage according to the 2009 TNM Staging system).
4. Patients who have not previously received systemic therapy, ECOG (Eastern Cooperative Oncology Group)≤2;
5. expected survival >3 months;
6. all patients signed informed consent.
7. blood routine indexes: neutrophils ≥1.5*109, platelets ≥100*109, hemoglobin ≥90g/L;
8. liver function: bilirubin ≤ normal upper limit 1.5 times, ALT/AST≤ normal upper limit 2.5 times;Serum creatinine ≤ 1.5 times of normal upper limit
9. the following diseases did not appear within 12 months: myocardial infarction, severe or unstable angina pectoris, asymptomatic heart failure, cardiovascular and cerebrovascular accident or transient ischemic attack, etc.

Exclusion Criteria:

1. other malignancies previously or at the same time that are different from the primary site or histology of the tumor assessed in this study, except cervical carcinoma in situ, basal-cell carcinoma that has been fully treated, superficial bladder tumor (Ta, Tis, T1) or other malignancies that occurred before the enrollment and have been cured for more than 3 years;
2. renal decompensation requires hemodialysis or peritoneal dialysis;
3. arrhythmia need anti-arrhythmic treatment, symptomatic coronary artery disease or myocardial ischemia (myocardial infarction), nearly six months, or congestive heart failure than NYHA Ⅱ level; Hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg) that has been treated with 2 or more antihypertensive treatments and still cannot be controlled;
4. severe active clinical infection;
5. patients with coagulation disorder or bleeding constitution;
6. major surgery or severe trauma was performed within 4 weeks before enrollment;
7. a history of allogeneic organ transplantation or bone marrow transplantation;
8. drug abuse and medical, psychological or social conditions that may interfere with patients' participation in research or affect the evaluation of results;
9. known or suspected allergy to the study drug;
10. those who received treatment other than this study within 4 weeks prior to and during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ORR per RECIST v1.1 and imRECIST as assessed by investigators | 3 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1 and imRECIST

SECONDARY OUTCOMES:
DCR per RECIST v1.1 and imRECIST as assessed by investigators | 3 years
  ORR is the proportion of subjects with complete response(CR), partial response(PR) or stable disease (SD) based on RECIST v1.1 and imRECIST
OS | 3 years
  OS is the time from the first use of a therapeutic drug to death from any cause
PFS per RECIST v1.1 and imRECIST as assessed by investigators | 3 years
  PFS is the time from the first use of a therapeutic drug to disease progression or death from any cause, progression is assessed by investigators based on RECIST v1.1 and imRECIST
Life quality Questionnaire composite | 3 years
  Evaluate life quality using EuroQol Five Dimensions Questionnaire (EQ-5D). EQ-5D included two aspects: EQ-5D Descriptive System and the EQ-5D visual analogue scale (EQ-VAS).
  In the description system, health status will be evaluated in 5 aspects: Mobility, Self-care, Usual Activities, Pain/Discomfort, Anxiety/Depression.
  EQ-VAS ranges from 0 to 100, higher scores indicate better health.
Pain score | 3 years
  Evaluate pain using visual analogue scale (VAS), range from 0 to 10, higher scores predict a poor prognosis.

OTHER OUTCOMES:
Treatment-related adverse events | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0, also types and degree

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zeng, Professor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol
Time Frame: Data would be available starting from the time when summary data are published or otherwise made available, for 3 years.
Access Criteria: Other researchers access the data by sending an email to our PI.

REFERENCES:
- [Background] Ljungberg B, Albiges L, Abu-Ghanem Y, Bedke J, Capitanio U, Dabestani S, Fernandez-Pello S, Giles RH, Hofmann F, Hora M, Klatte T, Kuusk T, Lam TB, Marconi L, Powles T, Tahbaz R, Volpe A, Bex A. European Association of Urology Guidelines on Renal Cell Carcinoma: The 2022 Update. Eur Urol. 2022 Oct;82(4):399-410. doi: 10.1016/j.eururo.2022.03.006. Epub 2022 Mar 26. PMID 35346519
- [Background] Diaz-Montero CM, Rini BI, Finke JH. The immunology of renal cell carcinoma. Nat Rev Nephrol. 2020 Dec;16(12):721-735. doi: 10.1038/s41581-020-0316-3. Epub 2020 Jul 30. PMID 32733094
- [Background] Motzer RJ, Tannir NM, McDermott DF, Aren Frontera O, Melichar B, Choueiri TK, Plimack ER, Barthelemy P, Porta C, George S, Powles T, Donskov F, Neiman V, Kollmannsberger CK, Salman P, Gurney H, Hawkins R, Ravaud A, Grimm MO, Bracarda S, Barrios CH, Tomita Y, Castellano D, Rini BI, Chen AC, Mekan S, McHenry MB, Wind-Rotolo M, Doan J, Sharma P, Hammers HJ, Escudier B; CheckMate 214 Investigators. Nivolumab plus Ipilimumab versus Sunitinib in Advanced Renal-Cell Carcinoma. N Engl J Med. 2018 Apr 5;378(14):1277-1290. doi: 10.1056/NEJMoa1712126. Epub 2018 Mar 21. PMID 29562145
- [Background] 2022 ASCO # Oral abstract 106.